CLINICAL TRIAL: NCT01621243
Title: A Phase I/II, Two-Part, Multicenter Study to Evaluate the Safety and Efficacy of M402 in Combination With Nab-Paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Brief Title: M402 in Combination With Nab-Paclitaxel and Gemcitabine in Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated after a pre-planned futility analyses showed an insufficient level of efficacy in the study population to warrant continuation.
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M402-103
Record Dates: First submitted 2012-05-22; First posted 2012-06-18 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: necuparanib; gemcitabine; heparin; low molecular weight heparin; nab-Paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nab-paclitaxel, gemcitabine, placebo (Placebo Comparator): Part A: Not applicable.
  Part B: nab-paclitaxel, gemcitabine, and placebo. Placebo administered daily along with nab-paclitaxel and gemcitabine administration on Day 1, Day 8, and Day 15 of each 28-day cycle.
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine; Drug: placebo
- nab-paclitaxel, gemcitabine, necuparanib (Experimental): Part A: Following a single-dose of necuparanib and a 7-day follow-up period, necuparanib was administered daily along with nab-paclitaxel and gemcitabine administration on Day 1, Day 8, and Day 15 of each 28-day cycle. Dose escalation of necuparanib proceeded by cohort in a 3+3 design.
  Part B: A fixed dose of necuparanib will be administered daily along with nab-paclitaxel and gemcitabine administration on Day 1, Day 8, and Day 15 of each 28-day cycle.
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine; Drug: Necuparanib

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel dosed on Day 1, Day 8, Day 15 of each 28-day cycle
  Other Names: Abraxane (nab-paclitaxel)
Drug: gemcitabine — gemcitabine will be dosed on Day 1, Day 8, Day 15 of each 28-day cycle
  Other Names: Gemzar (gemcitabine)
Drug: placebo — Placebo will be dosed daily
  Arms: nab-paclitaxel, gemcitabine, placebo
Drug: Necuparanib — Necuparanib will be dosed daily
  Arms: nab-paclitaxel, gemcitabine, necuparanib

SUMMARY:
People with primary metastatic pancreatic cancer will be treated with nab-paclitaxel and gemcitabine in combination with an investigational agent called necuparanib (M402). It is made from heparin, which is a well known blood thinner. Blood thinners have been shown in prior animal and human studies to have anti-cancer effects. Necuparanib has been re-engineered from heparin to have much lower blood thinning activity while keeping the anti-tumor activity. The investigators are testing whether necuparanib administered in combination with nab-paclitaxel and gemcitabine may be more effective than nab-paclitaxel and gemcitabine.

DETAILED DESCRIPTION:
Part A was an open-label, multiple ascending dose patient study of necuparanib given first as a single dose and then daily in combination with the nab-paclitaxel and gemcitabine regimen. It was conducted to evaluate the safety and tolerability of necuparanib alone and in combination with nab-paclitaxel and gemcitabine and to recommend a necuparanib dose regimen for subsequent evaluation in Part B. Part B is a randomized, double-blind study investigating the antitumor activity of necuparanib in combination with nab-paclitaxel and gemcitabine compared with nab-paclitaxel, gemcitabine, and placebo. In both Parts A and B, a treatment period consists of one 28-day cycle. The Study Patient and Investigator can decide to continue with additional 28-day cycles according to the patient's status at the end of each 28-day cycle. Part A has completed enrollment and Part B is currently open.

Part A - Primary Objectives:

* To evaluate the safety and tolerability of necuparanib in combination with nab-paclitaxel and gemcitabine.
* To determine the dose of necuparanib to be carried forward into Part B.

Part B - Primary Objective:

To evaluate overall survival in patients treated with necuparanib + nab-paclitaxel + gemcitabine compared with placebo + nab-paclitaxel + gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Confirmed pancreatic ductal adenocarcinoma
* Metastatic disease as documented by CT scan or MRI (locally advanced disease only NOT eligible)
* At least 1 site of disease measurable by RECIST ver1.1
* ECOG performance status of 0 to 1
* Adequate bone marrow, renal capacity and hepatic function
* Willing to administer daily subcutaneous injections at home

Exclusion Criteria:

* Any prior radiotherapy, chemotherapy, surgery, or investigational therapy for adjuvant or metastatic pancreatic cancer
* History of suspected history, or presence of heparin induced toxicity (w/ or w/o thrombosis)
* History of unexplained bleeding episodes within 3 months of M402 dosing
* Received thrombolytic agents w/in the previous month
* Had full-dose anticoagulation with heparin, enoxaparin, dalteparin, other LMWH, a/or other anticoagulants w/in 90 days before first dose of M402
* High cardiovascular risk, including but not limited to, recent coronary stenting or myocardial infarction in the past year
* Major trauma or surgery w/in prior 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-05; Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Part A: Safety | Part A: Baseline to 28 days after first-dose and end of study
  At baseline and then each of 6 visits after the start of dosing in a 28-day treatment cycle, adverse event surveillance, liver function enzyme levels, WBC with differential, ANC, aPTT, and PT are measured. This is repeated for each 28 day treatment cycle until disease progression or end of treatment. A final assessment is performed 30 days post-final necuparanib dose.
Part B: Overall Survival | Time in months from first dose of study medication until death
  Time in months from first dose of study medication until death

SECONDARY OUTCOMES:
Part A: Maximum concentration of necuparanib | Baseline to 28 days after first dose.
  One before and seven blood samples after the first dose followed by 5 additional lab draws, once at each of the 5 remaining visits in the first 28-day cycle.
Part B: Duration of progression-free survival | Time from first dose of study drug until disease progression
  Time in months from first dose of study drug until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: James Roach, MD, Study Director — Momenta Pharmaceuticals
Locations (37):
- United States (34):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Colorado School of Medicine - Division of Medical Oncology, Aurora, Colorado
  - Poudre Valley Health System, Fort Collins, Colorado
  - Hartford Healthcare Cancer Institute at Midstate Medical Center, Meriden, Connecticut
  - Florida Hospital Tampa, Tampa, Florida
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Crescent City Research Consortium, Marrero, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland- St Joseph's Medical Center, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota Community Clinical Oncology Program, Saint Louis Park, Minnesota
  - University of Kansas Cancer Center, Kansas City, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore-Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - Northwest Cancer Specialists, Portland, Oregon
  - Penn State Hershey Cancer Center, Hershey, Pennsylvania
  - Cancer Center of the Carolinas/ITOR, Greenville, South Carolina
  - University of Texas Health Sciences Center, San Antonio, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - Texas Oncology, Tyler, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (3):
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM Hospital St-Luc, Montreal, Quebec

REFERENCES:
- [Derived] O'Reilly EM, Barone D, Mahalingam D, Bekaii-Saab T, Shao SH, Wolf J, Rosano M, Krause S, Richards DA, Yu KH, Roach JM, Flaherty KT, Ryan DP. Randomised phase II trial of gemcitabine and nab-paclitaxel with necuparanib or placebo in untreated metastatic pancreas ductal adenocarcinoma. Eur J Cancer. 2020 Jun;132:112-121. doi: 10.1016/j.ejca.2020.03.005. Epub 2020 Apr 28. PMID 32361265
- [Derived] O'Reilly EM, Roach J, Miller P, Yu KH, Tjan C, Rosano M, Krause S, Avery W, Wolf J, Flaherty K, Nix D, Ryan DP. Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of Necuparanib Combined with Nab-Paclitaxel and Gemcitabine in Patients with Metastatic Pancreatic Cancer: Phase I Results. Oncologist. 2017 Dec;22(12):1429-e139. doi: 10.1634/theoncologist.2017-0472. Epub 2017 Nov 20. PMID 29158367